CLINICAL TRIAL: NCT01272440
Title: PEG-asparaginase Treatment in the NOPHO ALL-2008 Protocol: Antibody Formation, Pharmacokinetics, Pharmacodynamics and Side Effects.
Brief Title: A Drug Monitoring Study on PEG-asparaginase Treatment in Children Diagnosed Acute Lymphoblastic Leukaemia
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Louise Tram Henriksen, MD, Aarhus University Hospital
Other Study IDs: LTH-1
Record Dates: First submitted 2011-01-05; First posted 2011-01-07 (Estimated); Last update posted 2013-11-13 (Estimated); Status verified 2013-11

CONDITIONS: Acute Lymphoblastic Leukaemia
Keywords: PEG-asparaginase; children; pharmacokinetics; antibodies; acute lymphoblastic leukaemia; adverse effects
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, Cerebrospinal fluid
Oversight: Data Monitoring Committee: Yes

SUMMARY:
Asparaginase is an important drug i the treatment of childhood leukaemia.

The aim of this project is to study the pharmacokinetics, pharmacodynamics and antibody development and hypersensitivity reactions during prolonged PEG-asparaginase treatment.

Study part 1) Asparaginase pharmacokinetics and pharmacodynamics during prolonged PEG-asparaginase treatment: A NOPHO ALL-2008 study

Study part 2) Asparagine depletion in cerebrospinal fluid: A NOPHO ALL-2008 study

Study part 3) A characterization of PEG-asparaginase hypersensitivity in children treated according to the NOPHO ALL 2008 protocol

Perspectives: New knowledge about PEG-asparaginase treatment regarding dosing, dosing interval, adverse effects and EFS, which may lead to improved future therapy

Patients: Children diagnosed with acute lymphoblastic leukaemia in the Nordic Countries

ELIGIBILITY:
Inclusion Criteria:

Children aged between 1 and 18 years old, diagnosed ALL and treated according to the NOPHO-ALL 2008 protocol and who have accepted to participate in this study

Exclusion Criteria:

Children that does not attend the NOPHO-ALL 2008 protocol but receives standard treatment

Ages: 1 Year to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Children aged between 1 and 18 years old, diagnosed ALL and treated according to the NOPHO-ALL 2008 protocol
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2011-01; Primary Completion 2015-12 (Estimated); Study Completion 2015-12 (Estimated)

PRIMARY OUTCOMES:
Asparagine depletion | Up to 30 weeks of treatment
  Blood samples and cerebrospinal fluid samples are collected at certain timepoints during 30 weeks of treatment with PEG-asparaginase. They are analyzed for asparagine, asparaginase-enzyme activity and asparaginase-antibodies.These measures tell about the effect of the drug, PEG-asparaginase.

CONTACTS AND LOCATIONS:
Overall Officials: Louise T Henriksen, MD, Principal Investigator — Aarhus University Hospital
Locations (1):
- Paediatric department, Skejby University hospital, Aarhus, Denmark, Denmark